CLINICAL TRIAL: NCT01326559
Title: Phase II Study to Evaluate Induction Chemotherapy Using Docetaxel, Cisplatin and Fluorouracil Followed by Weekly Docetaxel and Cetuximab in Concurrence With Intensity-modulated Radiotherapy for Locally Recurrent Nasopharyngeal Carcinoma (NPC)
Brief Title: Study to Evaluate Induction Chemotherapy Using Docetaxel, Cisplatin and Fluorouracil in Concurrence With Intensity-modulated Radiotherapy for Local Recurrent Nasopharyngeal Carcinoma (NPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hong Kong Nasopharyngeal Cancer Study Group Limited (Other)
Collaborators: The University of Hong Kong (Other); Sanofi (Industry); Merck Sharp & Dohme LLC (Industry); Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Dr. ANNE W M LEE, Chief of Service, Dept of Clinical Oncology, PYNEH, Hong Kong Nasopharyngeal Cancer Study Group Limited
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-1001 trial
Record Dates: First submitted 2011-03-22; First posted 2011-03-31 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: induction chemotherapy; docetaxel; cisplatin; fluorouracil; cetuximab; intensity-modulated radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Docetaxel; Cisplatin; Fluorouracil; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental 1 (Experimental): Induction chemotherapy using Docetaxel, Cisplatin and 5-FU for week 1 to week 9 and followed by concurrent chemoradiation plus cetuximab from week 10 to week 16
  Interventions: Drug: Docetaxel, Cisplatin, 5-FU and Cetuximab

INTERVENTIONS:
Drug: Docetaxel, Cisplatin, 5-FU and Cetuximab — Induction phase (Weeks 1-9):
  Drug Docetaxel Docetaxel 75 mg/m2 IV, D1 every 3 weeks for 3 cycles
  Drug Cisplatin Cisplatin 75 mg/m2 IV, D1 every 3 weeks for 3 cycles
  Drug Fluorouracil Fluorouracil 750 mg/m2 IV, D1-4 every 3 weeks for 3 cycles
  Concurrent phase (weeks 10-16):
  Drug Docetaxel Docetaxel 15 mg/m2 IV, D1 weekly for 7 weeks (Weeks 10-16)
  Drug Cetuximab Cetuximab 400 mg m2 IV, D1 initial dose, then 250 mg/m2 weekly for 7 week (Weeks 10-16)
  IMRT (60 Gy to GTV or biological dose equivalent): 2 Gy/fraction/day, D1-5 per week, for 6 weeks (Weeks 11-16)

SUMMARY:
Study Objective:

Primary

1. To evaluate the complete response (CR) rate with induction chemotherapy using Docetaxel, Cisplatin and Fluorouracil(TPF) followed by Docetaxel plus Cetuximab (TC) in concurrence with intensity-modulated radiotherapy (IMRT).

Secondary

1. To determine the overall response rate.
2. To determine the locoregional and distant control rate
3. To determine the progression-free survival (PFS)
4. To determine the overall survival (OS)
5. To determine the safety of the induction chemotherapy and concurrent chemoradiation plus Cetuximab.

ELIGIBILITY:
Inclusion criteria:

* Recurrent T3N0-N1M0 NPC (by AJCC/UICC 6th edition) and at least 1 year from the end of last primary course of radiotherapy
* Age > 18 to < 70 years
* Performance status: < 1 by ECOG System (Appendix I)
* Adequate bone marrow & renal function
* Patients having Bilirubin =< 1.5 x ULN, ASAT & ALST=< 1.5 x ULN, Serum creatinine=< 1.25 x ULN and / or Creatinine clearance >= 60ml/min
* Patients having WBC >= 3x10e9/L, Neutrophils 1.8x10e9/L, Platelets >= 100 x10e9/L,Hemoglobin >=10g/dL
* Signed written informed consent
* Patients must have at least one measurable lesion

Exclusion Criteria:

* Use of investigational agent within the past 28 days
* Pre-treatment with an anti-EGFR drug
* Severe cardiac disease such as heart failure, coronary artery disease or myocardial infarction within the last 12 months
* History of severe pulmonary diseases
* Active infection or other systemic disease under poor control
* Uncontrolled chronic neuropathy
* Know grade 3 or 4 allergic reaction to any of the components of the treatment
* Estimated life expectancy is less than 3 months
* Pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-06; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Complete response rate | 5 years
  Complete response rate is defined as the proportion of subjects with disappearance of all target lesions after induction and concurrent therapies.

SECONDARY OUTCOMES:
Overall response rate | 5 years
  Defined as the proportion of subjects with best response (confirmed CR or PR) compared to the overall treated group.
Locoregional and distant control rate | 5 years
  Defined as the proportion of subjects with no local or nodal progression or recurrence and no distant disease progression or recurrence compared to the overall treated group.
Progression free survival | 5 years
  Defined as the time in months from first dose of cetuximab until PD is observed or death occurs due to any cause within 90 days after the last tumour assessment or first cetuximab dose.
Overall survival | 5 years
  Defined as the time in months from first dose of cetuximab to the date of death is observed. If subject has not died, the survival time will be censored on the last date the subject was known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Anne W.M., F.R.C.R.(HK), Principal Investigator — Department of Clinical Oncology, Pamela Youde Nethersole Eastern Hospital, Hong Kong
Locations (4):
- China (4):
  - Department of Clinical Oncology, Queen Mary Hospital(QMH), Hong Kong, Hong Kong
  - Department of Clinical Oncology, Queen Mary Hospital, Hong Kong
  - Department of Clinical Oncology, Tuen Mun Hospital (TMH), Hong Kong, Hong Kong
  - Department of Oncology, Princess Margaret Hospital, Hong Kong

REFERENCES:
- [Background] Fu KK, Newman H, Phillips TL. Treatment of locally recurrent carcinoma of the nasopharynx. Radiology. 1975 Nov;117(2):425-31. doi: 10.1148/117.2.425. PMID 170644
- [Background] Pryzant RM, Wendt CD, Delclos L, Peters LJ. Re-treatment of nasopharyngeal carcinoma in 53 patients. Int J Radiat Oncol Biol Phys. 1992;22(5):941-7. doi: 10.1016/0360-3016(92)90792-g. PMID 1555986
- [Background] Wang CC. Re-irradiation of recurrent nasopharyngeal carcinoma--treatment techniques and results. Int J Radiat Oncol Biol Phys. 1987 Jul;13(7):953-6. doi: 10.1016/0360-3016(87)90030-7. PMID 3597157
- [Background] Teo PM, Kwan WH, Chan AT, Lee WY, King WW, Mok CO. How successful is high-dose (> or = 60 Gy) reirradiation using mainly external beams in salvaging local failures of nasopharyngeal carcinoma? Int J Radiat Oncol Biol Phys. 1998 Mar 1;40(4):897-913. doi: 10.1016/s0360-3016(97)00854-7. PMID 9531376
- [Background] Leung TW, Tung SY, Sze WK, Sze WM, Wong VY, Wong CS, O SK. Salvage radiation therapy for locally recurrent nasopharyngeal carcinoma. Int J Radiat Oncol Biol Phys. 2000 Dec 1;48(5):1331-8. doi: 10.1016/s0360-3016(00)00776-8. PMID 11121630
- [Background] Poon D, Yap SP, Wong ZW, Cheung YB, Leong SS, Wee J, Tan T, Fong KW, Chua ET, Tan EH. Concurrent chemoradiotherapy in locoregionally recurrent nasopharyngeal carcinoma. Int J Radiat Oncol Biol Phys. 2004 Aug 1;59(5):1312-8. doi: 10.1016/j.ijrobp.2004.01.037. PMID 15275714
- [Background] Yan JH, Hu YH, Gu XZ. Radiation therapy of recurrent nasopharyngeal carcinoma. Report on 219 patients. Acta Radiol Oncol. 1983;22(1):23-8. doi: 10.3109/02841868309134335. PMID 6305129
- [Background] Lu TX, Mai WY, Teh BS, Zhao C, Han F, Huang Y, Deng XW, Lu LX, Huang SM, Zeng ZF, Lin CG, Lu HH, Chiu JK, Carpenter LS, Grant WH 3rd, Woo SY, Cui NJ, Butler EB. Initial experience using intensity-modulated radiotherapy for recurrent nasopharyngeal carcinoma. Int J Radiat Oncol Biol Phys. 2004 Mar 1;58(3):682-7. doi: 10.1016/S0360-3016(03)01508-6. PMID 14967420
- [Background] Chua DT, Sham JS, Leung LH, Au GK. Re-irradiation of nasopharyngeal carcinoma with intensity-modulated radiotherapy. Radiother Oncol. 2005 Dec;77(3):290-4. doi: 10.1016/j.radonc.2005.10.010. Epub 2005 Nov 8. PMID 16289398
- [Background] Chua DT, Sham JS, Au GK. Induction chemotherapy with cisplatin and gemcitabine followed by reirradiation for locally recurrent nasopharyngeal carcinoma. Am J Clin Oncol. 2005 Oct;28(5):464-71. doi: 10.1097/01.coc.0000180389.86104.68. PMID 16199985
- [Background] Vermorken JB, Remenar E, van Herpen C, Gorlia T, Mesia R, Degardin M, Stewart JS, Jelic S, Betka J, Preiss JH, van den Weyngaert D, Awada A, Cupissol D, Kienzer HR, Rey A, Desaunois I, Bernier J, Lefebvre JL; EORTC 24971/TAX 323 Study Group. Cisplatin, fluorouracil, and docetaxel in unresectable head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1695-704. doi: 10.1056/NEJMoa071028. PMID 17960012
- [Background] Bonner JA, Harari PM, Giralt J, Azarnia N, Shin DM, Cohen RB, Jones CU, Sur R, Raben D, Jassem J, Ove R, Kies MS, Baselga J, Youssoufian H, Amellal N, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for squamous-cell carcinoma of the head and neck. N Engl J Med. 2006 Feb 9;354(6):567-78. doi: 10.1056/NEJMoa053422. PMID 16467544
- [Background] Nakata E, Hunter N, Mason K, Fan Z, Ang KK, Milas L. C225 antiepidermal growth factor receptor antibody enhances the efficacy of docetaxel chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2004 Jul 15;59(4):1163-73. doi: 10.1016/j.ijrobp.2004.02.050. PMID 15234052
- [Background] Posner MR, Hershock DM, Blajman CR, Mickiewicz E, Winquist E, Gorbounova V, Tjulandin S, Shin DM, Cullen K, Ervin TJ, Murphy BA, Raez LE, Cohen RB, Spaulding M, Tishler RB, Roth B, Viroglio Rdel C, Venkatesan V, Romanov I, Agarwala S, Harter KW, Dugan M, Cmelak A, Markoe AM, Read PW, Steinbrenner L, Colevas AD, Norris CM Jr, Haddad RI; TAX 324 Study Group. Cisplatin and fluorouracil alone or with docetaxel in head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1705-15. doi: 10.1056/NEJMoa070956. PMID 17960013